CLINICAL TRIAL: NCT05665179
Title: Removing Barriers: Community Partnering for Innovative Solutions to the Opioid Crisis
Acronym: RB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Cordova, Associate Professor of Social Work, School of Social Work, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00152102
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Opioid Use Disorder; Alcohol Use Disorder; Health Risk Behaviors; Criminal Behavior; Housing Problems; Overdose of Opiate
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism; Health Risk Behaviors; Criminal Behavior; Opiate Overdose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Receives tutorial for free online legal resolution at treatment center
  Interventions: Behavioral: Removing Barriers to Recovery
- Control (No Intervention): The control group is not provided the experimental intervention.

INTERVENTIONS:
Behavioral: Removing Barriers to Recovery — Experimental patients are provided no-cost legal services in-person at addiction treatment centers using an online platform
  Arms: Treatment

SUMMARY:
The opioid epidemic has become one of America's deadliest crises, surpassing car crashes, firearms, and HIV/AIDS as a leading cause of death for Americans under fifty years of age. People trying to recover from opioid-use disorder face many obstacles. Obstacles such as minor legal problems (e.g., arrest warrants for failure to pay a fine, failure to appear in court, or late child support payments) can undermine the stability needed to overcome opioid dependence. Outstanding legal obligations make it difficult to find jobs and to secure housing. They can result in removal from treatment programs as well as incarceration. Resolving these legal problems requires coordination, organization, preparation, travel, and time-expectations that may be problematic for many people in the early stages of recovery. Technology has the potential to make resolving these legal problems much easier. Online platform technology is now available that can guide people in recovery through the resolution of many legal problems at no cost and without an attorney, potentially doing so quickly, remotely, and at any time of day.

This study of individuals in treatment in Michigan tests whether resolving outstanding legal issues improves drug treatment outcomes. The research also examines whether and to what extent resolving legal issues supports family reunification, reduces future criminal behavior, and improves access to jobs and housing for clients in treatment for opioid use disorder. A randomized controlled trial (RCT) is used to determine the effects of resolving legal issues on these outcomes. For identification, the investigators leverage the random assignment of legal services to treatment center clients, along with the random assignment of clients to treatment centers by birth month. We assemble a novel longitudinal dataset of hundreds of clients in treatment for substance use disorder and link these clients to several administrative datasets and qualitative data, which allows for measurement of: (1) substance use behaviors and (2) justice-system involvement, including civil and criminal legal system encounters. This study also uses linked client and administrative data to research the population in opioid treatment centers, follow-up behaviors, and whether the consequences of providing no-cost legal services differ by client background. Findings from this research will improve America's understanding of the acute socio-legal needs faced by those experiencing opioid use disorder and provide recommendations to help target resources toward the areas that best support long-term abstinence from opioids and other drugs.

ELIGIBILITY:
Inclusion Criteria:

*Receiving substance use disorder treatment services

Exclusion Criteria:

*Not receiving substance use disorder treatment services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-12-23 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of substance misuse | 1 year
  Consulting electronic medical records, we measure how frequently the participant report using substance(s). Daily rates will be recorded or calculated if frequency of use is recorded in weekly, monthly, or annual terms.
Quantity of substance(s) | 1 year
  Consulting electronic medical records, what is the mean quantity/measurement of substance(s) reported by participant per use. For alcohol, this is mean number of drinks per day(indicate beer, wine, liquor). For drugs this should be recorded in the standard measurement commonplace to that specific drug as recorded in the medical record, such as marijuana use in mean grams per day.

SECONDARY OUTCOMES:
Frequency of substance misuse | 2 years
  Consulting electronic medical records, we measure how frequently the participant report using substance(s). Daily rates will be recorded or calculated if frequency of use is recorded in weekly, monthly, or annual terms.
Quantity of substance(s) | 2 years
  Consulting electronic medical records, what is the mean quantity/measurement of substance(s) reported by participant per use. For alcohol, this is mean number of drinks per day(indicate beer, wine, liquor). For drugs this should be recorded in the standard measurement commonplace to that specific drug as recorded in the medical record, such as marijuana use in mean grams per day.
Count of justice system involvement | 1 year
  Utilizing State Court Administrative Office data, indicate count of all misdemeanor charges and count of felony charges. Using public records search on participant last known address, indicate count of civil case(s) including divorce, custody, eviction, bankruptcy, debt collection.
Justice system involvement case type | 1 year
  Utilizing State Court Administrative Office data, indicate case type of misdemeanor charges and count of felony charges. Using public records search on participant last known address, indicate case type of civil case(s) including divorce, custody, eviction, bankruptcy, debt collection.
Count of justice system involvement | 2 years
  Utilizing State Court Administrative Office data, indicate count of misdemeanor charges and count of felony charges. Using public records search on participant last known address, indicate count of civil case(s).
Case type of justice system involvement | 2 years
  Utilizing State Court Administrative Office data, indicate case type of all misdemeanor charges and count of felony charges. Using public records search on participant last known address, indicate case type of civil case(s) including divorce, custody, eviction, bankruptcy, debt collection.

CONTACTS AND LOCATIONS:
Overall Officials: David Cordva, PhD, Principal Investigator — Associate Professor
Locations (2):
- United States (2):
  - Home of New Vision, Ann Arbor, Michigan
  - Dawn Farm, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: Yes
deidentified data only
Supporting Information: Study Protocol, ICF
Time Frame: within 1 year of study completion and follow-up administrative data linkages complete
Access Criteria: public

REFERENCES:
- [Derived] O'Neil MM, Johnson RA, Cordova D, Pryor J, Pinals DA. A legal dispute resolution intervention for patients with substance use disorders: a study protocol for a randomized controlled trial. BMC Public Health. 2023 Mar 6;23(1):435. doi: 10.1186/s12889-023-15296-5. PMID 36879259